CLINICAL TRIAL: NCT03410238
Title: Translation of an Evidenced-Based Violence Intervention for Adolescents in Primary Care
Brief Title: Saferteens in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Maureen A Walton, Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00133654
Record Dates: First submitted 2018-01-18; First posted 2018-01-25 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants receive Saferteens Brief Intervention and a brochure containing psycho-education and resources.
  Interventions: Behavioral: Saferteens Brief Intervention
- Control (No Intervention): Participants receive a brochure containing psycho-education and resources only.

INTERVENTIONS:
Behavioral: Saferteens Brief Intervention — A 30 minute private one-on-one brief motivational interviewing intervention administered by clinic staff. The goal of the intervention is to reduce and prevent youth violence using techniques to change behavior in a respectful, non-confrontational, and non-judgmental manner. This one-on-one counseling approach emphasizes individual choice and responsibility and differentiates between future goals/values and current behavior. In the 2 months following the intervention, participants will receive booster text messages tailored to their responses during the intervention.
  Arms: Treatment

SUMMARY:
The SafERteens Study demonstrated the efficacy of a brief intervention (BI) for violence on changing attitudes, self-efficacy, and reducing violent behaviors, peer victimization, and violence-related consequences among adolescents in the emergency department (ED). Using a RE-AIM framework to measure outcomes (Reach, Effectiveness, Adoption, Implementation, and Maintenance), a study was conducted to translate this BI for violence into clinical practice in the ED. A SafERteens Implementation Package was created, which is housed on a website (www.saferteens.org), and includes: 1) a self-administered screen via iPad; 2) training materials (e.g., standardized patient videos); 3) clinician tools to guide intervention delivery; and 4) a tailored text message booster program.

To increase reach and impact on reducing youth violence, this project will implement SafERteens into primary care. Primary care represents a logical dissemination channel for the SafERteens intervention because 95% of adolescents report having a usual place for primary health care, with 75% receiving medical care in the past six months. Violence interventions have yet to be systematically implemented in primary care settings despite the alarming prevalence of violent behaviors among adolescents.

DETAILED DESCRIPTION:
This pilot study will customize the SafERteens intervention for the unique constraints of primary care settings and test implementation of the Saferteens brief intervention in primary care using the RE-AIM framework: reach (e.g., number of patients screened and given BI); effectiveness (e.g., change in violent behaviors, peer victimization, and violence-related consequences among intervention and control groups); adoption (e.g., number of providers trained, hours participated in training); implementation (e.g., participant ratings of intervention); and maintenance (e.g., ongoing screening and interventions during maintenance phase). Specifically, a control sample of youth ages 14-18 will be obtained, who will complete a baseline and 3-month follow-up survey, but who will not receive the intervention, and an intervention sample of youth ages 14-18 will be obtained, who will receive the Saferteens BI and will complete a baseline and 3-month follow-up survey. These data will provide a control sample for testing effectiveness of the Saferteens intervention package, versus the intervention sample.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (ages 14-18) presenting to primary care
* Screen positive for past year violent behavior (physical aggression) toward a friend, stranger, acquaintance, or dating partner (e.g., "have you pushed, hit, slapped, punched, kicked, been in a serious physical fight, group fight, or beat someone up

Exclusion Criteria:

* Adolescents who do not understand English
* Adolescents deemed unable to provide informed assent/consent (e.g., mental incompetence)

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Violent Behavior | 3 months post-baseline
  Change in violent behavior is assessed using 10 validated items from the National Longitudinal Study of Adolescent Health and Conflict Tactics Scale and assess the frequency of moderate (e.g., pushed or shoved) and severe (e.g., hit or punched, used a knife/gun) aggression towards peers. A composite score will be computed by summing the midpoint of responses to facilitate assessing change between baseline and follow-up.
Change in Victimization by peers | 3 months post-baseline
  Change in victimization by peers is assessed using 2 validated items from the Conflict Tactics Scale which assess the frequency of moderate and severe peer victimization. A composite score will be computed by summing the midpoint of the items to facilitate measuring change between baseline and follow-up.
Change in Violence Consequences | 3 months post-baseline
  Change in violence consequences is assessed using a 7 item scale. This scale was developed for the original SafERteens study and inquires about possible consequences of fighting, like trouble at school and expressed concern about fighting by family members or friends. A composite score will be computed to facilitate measuring change between baseline and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen A Walton, MPH, PHD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT03410238/ICF_000.pdf